CLINICAL TRIAL: NCT07027735
Title: Decellularized Human Placental Extracellular Matrix Tissue for Rotator Cuff Repair Augmentation
Acronym: ECMRCR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: CTM Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAV5510
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Standard Rotator Cuff Repair + Receives Allograft Treatment
  Interventions: Other: Rotator Cuff Repair with Allograft Patch
- Control Arm (Other): Standard Rotator Cuff Repair + NO Allograft Treatment
  Interventions: Other: Rotator Cuff Repair with No Augmentation

INTERVENTIONS:
Other: Rotator Cuff Repair with Allograft Patch — Rotator cuff repairs will be augmented with use of a decellularized human placental allograft patch
  Arms: Treatment Arm
Other: Rotator Cuff Repair with No Augmentation — Standard rotator cuff repair with no augmentation
  Arms: Control Arm

SUMMARY:
The rotator cuff is a set of muscles and tendons that help move the shoulder. Tears in the rotator cuff are common, particularly as people age. Consequently, rotator cuff repair surgeries are common, as well. Despite the frequency with which rotator cuff repairs are performed, there remains a high rate of postoperative failure to heal. In such situations, there is a lack of connective tissue establishment between the rotator cuff tendon and the bone. One strategy to attempt to improve healing of the rotator cuff tendon back to the bone is via the use of extracellular matrix allograft. This treatment is composed of tissue from other humans, which is stripped of its cells so that just the scaffolding around the cells remains. This decellularized scaffolding can be placed at the rotator cuff healing site in an attempt to augment healing. Both animal studies and human studies have shown promise with this approach. Of those patients enrolling in the study, 50% will be assigned at random to receive a standard rotator cuff repair AND allograft treatment, while 50% will be assigned at random to receive standard rotator cuff repair WITHOUT allograft treatment. All patients enrolled in the study will also obtain an MRI at one year following surgery in order to assess tendon healing. Of note, one-year postoperative MRIs are not standard following rotator cuff repair - only those enrolled in the study will receive this MRI. There will be no financial consequence of receiving this MRI.

DETAILED DESCRIPTION:
Rotator cuff repair is one of the most commonly performed orthopedic surgeries, with over 450,000 surgeries performed every year in the United States. Unfortunately, the failure rate postoperatively remains unacceptably high despite advances in surgical techniques and rehabilitation strategies. Clinical studies have shown that only about half of repaired rotator cuffs heal by 12 months following surgery, with the rate of recurrent tears ranging from 20% in the best case and as high as 94% in certain patient populations with massive tears. Animal model studies indicate that the high failure rate after surgical repair is due to a lack of regeneration of the native tendon-to-bone transitional tissue. This native transition zone, the enthesis, is a functionally graded mineralized fibrocartilaginous structure that minimizes stress concentrations at the interface between the mechanically dissimilar tissues of tendon and bone. Rather than re-formation of this fibrocartilaginous transition, necessary for effective load transfer between tendon and bone, an abrupt transition of fibrovascular scar forms at the healing interface and the underlying bone resorbs. remodeling and are used to augment the body's natural healing response. The efficacy of decellularized ECM treatment in rotator cuff repair, specifically, has been demonstrated by animal studies, which have shown that decellularized ECM contributes to cell ingrowth, improved remodeling, and, ultimately, an improved repair as gauged by biomechanical testing. Similarly, human studies have also been promising. Decellularized ECM treatment was shown to both reduce retear rate and improve patient outcome scores when used in the treatment of large to massive rotator cuff tears in humans.

Connective tissue is the fibrous extracellular matrix (ECM) that provides the physical structure and support of the body's tissues. The efficacy of decellularized ECMs to augment damaged tissue and support tissue repair throughout the body (e.g. tendon, ligament, bone, mucosal, and integumental) has been well-documented in the literature. Decellularized ECMs contain ECM components to support tissue remodeling and are used to augment the body's natural healing response. The efficacy of decellularized ECM treatment in rotator cuff repair, specifically, has been demonstrated by animal studies, which have shown that decellularized ECM contributes to cell ingrowth, improved remodeling, and, ultimately, an improved repair as gauged by biomechanical testing. Similarly, human studies have also been promising. Decellularized ECM treatment was shown to both reduce retear rate and improve patient outcome scores when used in the treatment of large to massive rotator cuff tears in humans.

This is a single center prospective randomized controlled trial. Subjects will be recruited from patients seen by one of three participating shoulder and elbow surgeons at outpatient visits for their rotator cuff tear diagnosis at Columbia University Medical Center or any of the affiliated hospitals and/or outpatient office spaces. Adult patients (age 18 years or older) with a diagnosis of full thickness rotator cuff tear who meet operative criteria, including significant pain and weakness that have failed nonoperative management or arose from an acute injury, will be included in this study. Patients with partial thickness tears, full thickness subscapularis tears, Goutallier grade 3 and 4 fatty degeneration, and/or prior rotator cuff surgeries will be excluded from the study. Patients will receive preoperative clearance in accordance with current practices. Post-transplant patients will receive screening for infectious diseases, including HIV, HBV, and HCV, prior to surgery. Patients will be randomized via simple randomization into one of two groups - standard arthroscopic repair with decellularized ECM vs. standard arthroscopic repair without decellularized ECM. Patients will be seen postoperatively at 2 weeks, 3 months, 6 months, and 12 months. All patients will undergo comparable rehabilitation programs. An MRI will be performed at 12 months postoperatively. Any incidental MRI findings will be dealt with in accordance with standard practice. The primary outcome measure will be the postoperative retear rate, measured on one year postoperative MRI. Secondary outcome measures will both additional MRI measurements, including tendon structural continuity and tendon thickness, as well as patient reported outcomes, including Constant-Murley score, American Shoulder and Elbow Surgeons score, VAS Pain scores, and EQ-5D-5L. Patient reported outcomes will be collected at all patient visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of full thickness rotator cuff tear

Exclusion Criteria:

* Partial thickness tears
* Full thickness subscapularis tears
* Goutallier grades 3 and 4
* Prior rotator cuff surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Retear Rate | 1 year
  The primary outcome measure will be the postoperative retear rate, measured on one-year postoperative MRI

SECONDARY OUTCOMES:
Tendon Structural Continuity (MRI) | 1 year
  MRI Measurement of Tendon Structural Continuity
Tendon Thickness (MRI) | 1 year
  MRI measurement of tendon thickness
Constant-Murley score | 1 year
  The Constant-Murley score is a 100-point scale used to assess shoulder function, with a higher score indicating better function. The components include Pain (0 - 15 points), Activities of Daily Living (0 - 20 points), Range of Motion (0 - 40 points), and Strength (0 -25 points). The full score range is 0 to 100.
American Shoulder and Elbow Surgeons (ASES) score | 1 year
  The American Shoulder and Elbow Surgeons (ASES) score is a patient-reported assessment of shoulder pain and function. It ranges from 0 to 100, with higher scores indicating better function. The ASES score combines a pain component (assessed using a Visual Analogue Scale (VAS) that ranges from 0 - 50) and a functional component (10 items, 5 points each). The full score range is 0 to 100.
Visual Analogue Scale (VAS) Pain scores | 1 year
  The VAS Pain full range is 0 to 10, with a higher score indicating worse pain imaginable.
EQ-5D Index Value (Utility Score) | 1 year
  The EQ-5D Index Value is a single number that summarizes the health state described by the EQ-5D questionnaire. The full range is 0 (worst health state, equivalent to death) to 1 (perfect health).
EuroQol Visual Analogue Scale (EQ VAS) | 1 year
  EQ-VAS is a self-reported measure used to assess a patient's health-related quality of life on a scale from 0 to 100. The scale ranges from "worst imaginable health" (0) to "best imaginable health" (100).

CONTACTS AND LOCATIONS:
Overall Officials: William Levine, MD, Principal Investigator — Columbia University
Locations (1):
- NewYorkPresbyterian Hospital @ Columbia, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No